CLINICAL TRIAL: NCT02979106
Title: Are Heterozygous Carriers for Hereditary Fructose Intolerance Predisposed to Metabolic Disturbances When Exposed to Fructose?
Brief Title: Metabolic Consequences of Heterozygous Hereditary Fructose Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor, University of Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PB_2016-00289 (302/14)
Record Dates: First submitted 2016-11-14; First posted 2016-12-01 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Hereditary Fructose Intolerance; Fructose Metabolism, Inborn Errors; Glucose Metabolism Disorders
MeSH Terms: conditions — Fructose Intolerance; Fructose Metabolism, Inborn Errors; Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oral fructose load (Experimental): test meal calculated to provide 25% of basal energy requirement containing 13C-labeled fructose (0.35 g/kg), protein (0.21 g/kg) and lipid (0.22 g/kg).
  Interventions: Other: Test meal

INTERVENTIONS:
Other: Test meal — Assessment of postprandial responses to a mixed meal containing fructose in carriers of one mutated ALDOB allele.

SUMMARY:
Background: High fructose intake increases blood lactate, triglyceride and uric acid concentrations. Uric acid may contribute to insulin resistance and dyslipidemia in the general population. In patients with hereditary fructose intolerance fructose consumption is associated with acute hypoglycemia, renal tubular acidosis, and hyperuricemia.

Objective: We investigated whether asymptomatic carriers for hereditary fructose intolerance (HFI) would have a higher sensitivity to adverse effects of fructose than the general population.

Design: Eight subjects heterozygous for HFI (hHFI; 4 males, 4 females) and eight controls received for 7 days a low fructose diet and on the eighth day ingested a test meal calculated to provide 25% of basal energy requirement containing labeled fructose (13C fructose 0.35 g/kg), protein (0.21 g/kg) and lipid (0.22 g/kg). Total fructose oxidation, total endogenous glucose production (by 6,6-2H2-glucose dilution), carbohydrate and lipid oxidation, lipids, uric acid, lactate, creatinine, urea and amino acids were monitored for 6 hours.

ELIGIBILITY:
Inclusion Criteria:

* 8 healthy Volunteers (4 male, 4 female) parents of a child with hereditary fructose intolerance with ALDOB with heterozygous mutation of ALDOB gene
* 8 healthy Volunteers (4 male, 4 female), healthy with no mutation of ALDOB gene

Exclusion Criteria:

* Fasting glycemia > 7.0 mmol/L
* Fasting total triglycerides > 4.0 mmol/L
* Chronic renal insufficiency (eGFR ≤ 50 ml/min)
* Anemia (ferritin < 20 ug/L, hemoglobin < 13.5 ou 12.5 g/dl)
* Drugs
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Plasma glucose kinetics | -120 min before ingestion of a test meal to 360 min after ingestion of a test meal
  Modelling of rate of glucose appearance after administration of a bolus of 6,6-2H2 glucose (bolus, 2 mg/kg and continuous infusion, 0.02 mg/kg/min) will be measured in fasted and fed conditions

SECONDARY OUTCOMES:
Energy expenditure rate | 120 min before ingestion of a test meal, and every 30 min until 360 min after ingestion of a test meal
  Energy expenditure is measured by indirect calorimetry in fasted and fed conditions
Glucose oxidation rate | 120 min before ingestion of a test meal, and every 30 min until 360 min after ingestion of a test meal
  glucose oxidation is measured by indirect calorimetry in fasted and fed conditions
Plasma glucose concentration | -120 min before ingestion of a test meal, and every 30 min until 360 min after ingestion of a test meal
  plasma glucose concentration measured by glucose oxidase
plasma insulin concentration | -120 min before ingestion of a test meal, and every 30 min until 360 min after ingestion of a test meal
  Plasma insulin concentration measured by ELISA
Fructose oxidation | Every 30 min until 360 min after ingestion of a test meal
  Fructose oxidation is measured from 13CO2 production

CONTACTS AND LOCATIONS:
Overall Officials: Tappy Luc, MD, Study Director — University of Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Debray FG, Damjanovic K, Rosset R, Mittaz-Crettol L, Roux C, Braissant O, Barbey F, Bonafe L, De Bandt JP, Tappy L, Paquot N, Tran C. Are heterozygous carriers for hereditary fructose intolerance predisposed to metabolic disturbances when exposed to fructose? Am J Clin Nutr. 2018 Aug 1;108(2):292-299. doi: 10.1093/ajcn/nqy092. PMID 29955837